CLINICAL TRIAL: NCT02095379
Title: Oligosecretary Myeloma: Prevalence and Its Clinical Significance
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Kihyun Kim, Professor, Samsung Medical Center
Other Study IDs: 2014-02-055
Record Dates: First submitted 2014-02-13; First posted 2014-03-24 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-03

CONDITIONS: Multiple Myeloma
Keywords: oligosecretary multiple myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- oligosecretary: Multiple myeloma (MM) characterized by low levels of serum and urine monoclonal (M) protein below thresholds of measurable disease (a serum M protein ≥ 1g/dL, a urine M protein ≥ 200mg/day)
  Interventions: Other: oligosecretary

INTERVENTIONS:
Other: oligosecretary — not abvailable

SUMMARY:
In this study, the investigators aim to investigate the prevalence and clinical course of oligosecretary myeloma.

DETAILED DESCRIPTION:
Oligosecretary myeloma is a subgroup of multiple myeloma (MM) characterized by low levels of serum and urine monoclonal (M) protein below thresholds of measurable disease (a serum M protein ≥ 1g/dL, a urine M protein ≥ 200mg/day). Patients with oligosecretary myeloma do not have established methods for disease monitoring and clinical informations regarding oligosecretary myeloma are still largely unknown.

In this study, we aimed to investigate the prevalence and clinical course of oligosecretary myeloma.

ELIGIBILITY:
Inclusion Criteria:

* a subgroup of multiple myeloma (MM) characterized by low levels of serum and urine monoclonal (M) protein below thresholds of measurable disease (a serum M protein ≥ 1g/dL, a urine M protein ≥ 200mg/day)
* available clinical data

Exclusion Criteria:

* patients without available clinical data

Ages: 17 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: a subgroup of multiple myeloma (MM) characterized by low levels of serum and urine monoclonal (M) protein below thresholds of measurable disease (a serum M protein ≥ 1g/dL, a urine M protein ≥ 200mg/day)
Sampling Method: Non-Probability Sample
Enrollment: 390 (Actual)
Dates: Start 2013-10; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Number of patients with oligosecretary myeloma among multiple myeloma patients | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kihyun Kim, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea